CLINICAL TRIAL: NCT06638320
Title: Hepatitis Delta Virus Infection: Cross-sectional Study in Patients With Chronic Hepatitis B Virus Infection
Status: Active, not recruiting | Type: Observational
Sponsor: Tam Anh Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: TA0001
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-03

CONDITIONS: Hepatitis Delta With Hepatitis B Carrier State; Chronic Hepatitis b
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with chronic hepatitis B virus infection

SUMMARY:
The goal of this observational study is to determine the prevalence of hepatitis D virus (HDV) and the distribution of the HDV genotype in patients with chronic hepatitis B infection. It will also identify factors related to hepatitis D virus infection, such as characteristics of the study sample, vaccination history, drug use affecting hepatitis, family factors, environment, and lifestyle.

This study will be conducted at Tam Anh General Hospital, Bach Mai Hospital and Tam Anh TP. Ho Chi Minh General Hospital.

Participants will be interviewed directly through a questionnaire to collect some information related to epidemiological risk factors. A blood sample will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 16 years old undergo testing at the Testing Center of Tam Anh General Hospital or Tam Anh TP. Ho Chi Minh General Hospital, with chronic hepatitis B HBsAg (+) standards for six months or over or HBsAg (+) combined with HBcAb total (+) and HBcAb-immunoglobulin M (-).
* Patients ≥ 16 years old with chronic hepatitis B come to be examined or are inpatients at the Gastroenterology - Hepatobiliary Center of Bach Mai Hospital, diagnosed with hepatocellular carcinoma, and cirrhosis

Exclusion Criteria:

* Patients do not agree to participate in the study or refuse to sign a written informed consent.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients ≥ 16 years old with chronic hepatitis B, with hepatocellular carcinoma and cirrhosis or not, should be examined and treated at the Gastroenterology - Hepatobiliary Center of Bach Mai Hospital, Tam Anh General Hospital and Tam Anh TP. Ho Chi Minh General Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 2452 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of hepatitis D virus (HDV) in patients with chronic hepatitis B infection | Day 0 after recruitment
  The method of estimating prevalence based on the assumption of binary distribution will be applied to the entire study sample and each subgroup. The prevalence rate will be estimated by dividing the number of positive cases by the sample size. The 95% confidence interval of the prevalence will be calculated based on the binary distribution assumption. Prevalence will be estimated for each sex, age, and disease group (chronic hepatitis B, chronic hepatitis B with hepatocellular carcinoma, and cirrhosis).

SECONDARY OUTCOMES:
Distribution of the HDV genotype in patients with chronic hepatitis B infection | Day 0 after recruitment
  Testing for differences in genotypic distribution between disease groups will be analyzed using the Chi-squared test. The difference is statistically significant with p < 0.05.
Factors related to hepatitis D virus infection | Day 0 after recruitment
  The determination of the association between risk factors and HDV will be analyzed across the total study sample. The multivariate logistic regression method will be applied in determining the variables related to the probability of HDV infection. In this analysis, HDV infection (positive or negative) is the dependent variable; Independent variables include factors that reflect demography, lifestyle, environment, occupation, clinical history (including vaccinations), and history of drug use. There are many independent variables and these variables can be correlated, determining which one affects HDV infection is a major challenge. To solve this problem, we will apply the Bayesian Model Averaging method in the R library. Based on the results of this analysis, a prognostic model of the risk of HDV infection will be established.

CONTACTS AND LOCATIONS:
Locations (1):
- VNVC Tan Phu, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No